CLINICAL TRIAL: NCT02905409
Title: A Randomized, Double-masked, Multicenter, Controlled Study of Effects of Internal Membrane Peeling Surgery in Patients With Idiopathic Macular Hole Measured by Optical Coherence Tomography.
Brief Title: Study of Surgery in Patients With Idiopathic Macular Hole
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Beijing Hospital (Other Government); Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Mingwei Zhao, Head of Opthalmology Department, Principal Investigator, Clinical Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ILMIMH-CHINA
Record Dates: First submitted 2016-09-02; First posted 2016-09-19 (Estimated); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Idiopathic Macular Hole; Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 4PD diameter of ILM peeling in surgery (Active Comparator): Patients were stratified according to the macular hole closure index(MHCI) measured by OCT into 3 subgroup (MHCI<0.5, 0.5≤MHCI<0.7, MHCI≥0.7 ). And then randomized into 2 different intervention groups. If randomized into 4PD (papillary diameter) group, patients were given 4PD diameter of ILM (internal limiting membrane) peeling in surgery.
  Interventions: Procedure: ILM peeling surgery
- 2PD diameter of ILM peeling in surgery (Experimental): Patients were stratified according to the macular hole closure index(MHCI) measured by OCT into 3 subgroup (MHCI<0.5, 0.5≤MHCI<0.7, MHCI≥0.7 ). And then randomized into 2 different intervention groups. If randomized into 2PD (papillary diameter) group, patients were given 2PD diameter of ILM (internal limiting membrane) peeling in surgery.
  Interventions: Procedure: ILM peeling surgery

INTERVENTIONS:
Procedure: ILM peeling surgery — 4PD or 2PD diameter of ILM peeling in surgery was given to patients with IMH (idiopathic macular hole)

SUMMARY:
The purpose of this study is to determine the effects of two different internal limiting membrane peeling with distinct diameters after macular hole surgery on anatomical closure grades.

DETAILED DESCRIPTION:
The purpose of this study is to investigate two distinct diameter of internal limiting membrane peeling on anatomical outcomes of macular hole surgery with different preoperative idiopathic macular hole.

ELIGIBILITY:
Inclusion Criteria:

* patients with IMH
* patients signed the ICF
* patients with course of IMH less than 3 years

Exclusion Criteria:

* patients with hyper myopia
* patients with traumatic macular hole
* accompanied or secondary of other fundus disease
* open or reopen after receiving MH surgery
* patients with retinal detachment
* received vitrectomy due to other diseases
* glaucoma cannot be controled by medication
* patients with other retinal or choroidal disease that may affect VA
* poor patients compliance
* poor condition that cannot undertake the surgery
* dioptric media opacities which make it difficult to exam fundus or measure on OCT

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2016-08-31 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Anatomical closure grades in OCT | 6 months
  The anatomical outcomes were defined as good closure and poor closure.
Change of anatomical closure grades in OCT | 1 month, 3 months, 6 months, 1 year
  The anatomical outcomes were defined as good closure and poor closure.

SECONDARY OUTCOMES:
Change from baseline in BCVA (best corrected visual acuity). | 1 month, 3 months, 6 months, 1 year
  BCVA were measured by ETDRS chart.

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei Zhao, M.D, Study Director — Peking University People's Hospital; Hong Dai, M.D, Principal Investigator — Peking Union Medical College; Wenbin Wei, M.D, Principal Investigator — Beijing Tongren Hospital of Capital Medical University; Youxin Chen, M.D, Principal Investigator — Peking Union Medical College
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China